CLINICAL TRIAL: NCT03282357
Title: Evaluation of the Effectiveness and Safety of Radiesse for the Correction of Nasolabial Folds
Brief Title: Evaluation of the Effectiveness and Safety of Radiesse for the Correction of Nasolabial Folds in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: M900311004
Record Dates: First submitted 2017-09-12; First posted 2017-09-13 (Actual); Results first posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2020-11

CONDITIONS: Correction of the Moderate to Severe Nasolabial Folds

STUDY DESIGN:
Intervention Model Description: Split-face
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Radiesse (Experimental): Subjects are randomized as to which of the two nasolabial folds is treated with Radiesse.
  Interventions: Device: Radiesse injectable implant (dermal filler); Device: Restylane injectable implant (dermal filler)
- Restylane (Active Comparator): Subjects are randomized as to which of the two nasolabial folds is treated with Restylane.
  Interventions: Device: Radiesse injectable implant (dermal filler); Device: Restylane injectable implant (dermal filler)

INTERVENTIONS:
Device: Radiesse injectable implant (dermal filler) — Subdermal injection.
  Other Names: Calcium hydroxylapatite particles suspected in an aqueous based gel carrier.
Device: Restylane injectable implant (dermal filler) — Subdermal injection
  Other Names: Hyaluronic acid

SUMMARY:
The objectives of this study are to evaluate the effectiveness and safety of Radiesse for the correction of nasolabial folds (NLFs).

ELIGIBILITY:
Inclusion Criteria:

1. Is 22 - 65 years of age.
2. Has symmetrical NLFs of moderate or severe intensity (grade 3 or 4) on the WSRS as determined by the independent blinded evaluator and confirmed by the treating investigator at baseline.
3. Both folds must have the same NLF score at baseline. 4. Has signed an informed consent.

5. Understands and accepts the obligation not to receive any other facial procedures below the eyes during the study.

6. Understands and accepts the obligation to present for all scheduled follow-up visits and is logistically able to meet all study requirements.

7. Subjects of childbearing potential must have a negative pregnancy test result and must not be lactating at the Screening/Baseline Visit and be willing and able to use an acceptable method of birth control (e.g. barrier methods used with a spermicidal agent, hormonal methods, IUD, surgical sterilization, abstinence) during the study. Women will be considered if one of the following conditions is documented on the medical history:

1. Postmenopausal with last menstrual bleeding at least 12 months prior to study; and
2. Without a uterus and/or both ovaries.

Exclusion Criteria:

1. Has received surgical permanent implants, grafting, or surgery below the eyes on the face prior to injection or lower lid blepharoplasty within 6 months prior to injection.
2. Has received within the specified (washout) period or plans to receive treatment during the study conduct with a non-permanent facial filler in any facial area below the eyes:

   1. 12 months prior to study start - hyaluronic acid [HA] or collagen
   2. 18 months prior to study start - calcium hydroxylapatite [CaHA]
3. Has received at any time or plans to receive during the study a permanent facial filler (e.g. poly L-lactic acid [PLLA], polymethyl-methacrylate [PMMA], silicone) below the eyes.
4. Has received within the past 6 months or plans to receive during the study facial dermal resurfacing procedures (e.g. chemical peel, dermabrasion, ablative laser resurfacing), non-invasive skin-tightening (e.g. Thermage), botulinum toxin injections, mesotherapy, or fat injections below the eyes.
5. Has received in the past 2 weeks or plans to receive during the study any prescription wrinkle therapies (e.g. RENOVAÒ), topical steroids, skin irritating topical preparations, or pigmenting agents (self-tanning agents) for use on the face.
6. Has received in the past 2 months, or plans to receive immunosuppressive medications or systemic steroids (intranasal/inhaled steroids acceptable) during the study.
7. Has an acute inflammatory process or infection, active herpes infection, or history of chronic or recurrent infection or inflammation with the potential to interfere with the study results or increase the risk of adverse events (AEs).
8. Has a known bleeding disorder or has received or is planning to receive anti-coagulation, anti-platelet, or thrombolytic medications (e.g., warfarin), anti-inflammatory drugs (oral/injectable corticosteroids or NSAIDs (e.g., aspirin, ibuprofen), or other substances known to increase coagulation time (vitamins or herbal supplements, e.g., Vitamin E, garlic, gingko), from 10 days before injection to 3 days after injection.
9. Has a history of known liver or renal function disease/disorder or has clinically significant laboratory values at baseline.
10. Has a known history of allergic/anaphylactic reactions, including hypersensitivity to lidocaine or anesthetics of the amide type, or any of the device components.
11. Has a history of hyper- or hypo-pigmentation in the NLFs, keloid formation, or hypertrophic scarring.
12. Has recently lost or has the intention to lose a significant amount of weight ≥ 2 Body Mass Index (BMI) units during the course of the study.
13. Has any other medical condition with the potential to interfere with the study's conduct or assessments, or increase the risk of AEs.
14. Has participated in a study in the last 30 days or is enrolled or plans to enroll in any other interfering investigational study during participation in the study.
15. Is an employee or direct relative of an employee of the investigational department in site or the sponsor.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz North America, Inc.
Locations (4):
- China (4):
  - Peking University First Hospital, Merz Investigational Site #0860003, Beijing
  - Southern Medical University, Nanfang Hospital, Merz Investigational Site #0860006, Guangzhou
  - Zhejiang Provincial People's Hospital, Merz Investigational Site #0860005, Hangzhou
  - Xiangya Hospital Central South University, Department of Aesthetic Plastic Surgery, Merz Investigational Site #'0860007, Hunan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 4 investigative sites in China.
Pre-assignment Details: A total of 195 participants were screened, out of which 181 were randomized. Of these, 176 participants were treated and 164 participants completed the study.
Groups:
- Radiesse and Restylane: Participants received split-face nasolabial fold (NLF) treatment with study product Radiesse, subdermal injection, in one of the two NLFs and control product Restylane, subdermal injection, in the contralateral NLF on Day 1. Participants received an optional touch-up injection in one or both the NLFs at Month 1.
Period: Overall Study
Arm/Group | Radiesse and Restylane
Started | 181
Safety Evaluation Set | 176
Completed | 164
Not Completed | 17
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 4
Not completed — Adverse Event | 1
Not completed — Other | 9

BASELINE CHARACTERISTICS:
Population: The safety evaluation set (SES) was defined as all participants who received an investigational product.
Groups:
- Radiesse and Restylane: Participants received split-face NLF treatment with study product Radiesse, subdermal injection, in one of the two NLFs and control product Restylane, subdermal injection, in the contralateral NLF on Day 1. Participants received an optional touch-up injection in one or both the NLFs at Month 1.
Arm/Group | Radiesse and Restylane
Number analyzed (Participants) | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 170
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Han Chinese | 173
  Ethnicity: Other | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race (Asian) | 176
Region of Enrollment [Count of Participants; unit: Participants]
  China | 176
Fitzpatrick skin type [Count of Participants; unit: Participants] — Skin type I = white; very fair, red or blonde hair blue eyes; freckles; always burns, never tans, skin type II = white, fair, red or blond hair; blue, hazel or green eyes; usually burns, tans with difficulty, skin type III = cream white; fair with any eye or hair color (common); sometimes mild burn, gradually tans, skin type IV = brown; typical Mediterranean Caucasian skin; rarely burns, tans with ease, skin type V = dark brown; mid-eastern skin types; very rarely burns, tans easily, and skin type VI = black; never burns, tans very easily.
  Participants
    Type I | 0
    Type II | 0
    Type III | 147
    Type IV | 29
    Type V | 0
    Type VI | 0
    Missing | 0
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 159.9 (5.60)
Weight [Mean (Standard Deviation); unit: kilogram (Kg)] | 56.15 (8.434)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 21.87 (2.817)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of NLFs With Treatment Success at Month 6
Description: Treatment success was defined as a greater than or equal to (>=) 1-point improvement from baseline, as assessed by a blinded evaluator wrinkle severity rating scale (WSRS) scale. WSRS is a 5 point scale with scores as Score 1: Absent; Score 2: Mild; Score 3: Moderate; Score 4: Severe; Score 5: Extreme.
Time Frame: Month 6
Population: The per protocol set (PPS) was the subset of the full analysis set (FAS) without any major protocol deviations. The FAS was all participants randomized who received an investigational product with at least one post-baseline effectiveness assessment (WSRS, blind evaluator's Global Aesthetic Improvement Scale [GAIS] or participant's GAIS assessment).
Measure: Number; unit: Percentage of successfully treated NFLs
Units Other Than Participants: Nasolabial fold (NLF)
Groups:
- Radiesse: All participants received NLF treatment with study product Radiesse, subdermal injection, in one of the two NLFs on Day 1. Participants received an optional touch-up injection in the same NLF at Month 1.
- Restylane: All participants received NLF treatment with control product Restylane, subdermal injection, in the contralateral NLF on Day 1. Participants received an optional touch-up injection in the same NLFs at Month 1.
Arm/Group | Radiesse | Restylane
Number analyzed (Participants) | 171 | 171
Number analyzed (Nasolabial fold (NLF)) | 171 | 171
Percentage of successfully treated NFLs | 66.0 | 72.8
Statistical Analysis 1: Comparison: Radiesse vs Restylane; Test type: Non-Inferiority — Non-inferiority margin, delta = 10 percent (%). The two-sided 95% confidence interval (CI) for the differences between percentages was constructed using the Newcombe's recommended method; Difference in Percentage = -6.8, 95% CI 2-sided [-13.1 to -0.5]

2. Secondary Outcome: Percentage of NLFs With an Improvement in the Blinded Evaluator's GAIS Score at Month 6
Description: The blinded evaluator rated the current cosmetic result for each NLF according to the GAIS based on live assessments during the visit compared with photographs taken at baseline before administration of treatment on each NLF. An improvement on the GAIS was classified as "improved", "much improved", or "very much improved. The GAIS is a 7-point scale, where: +3 (very much improved), +2 (much improved), +1 (improved), 0 (no change), -1 (worse), -2 (much worse), and -3 (very much worse).
Time Frame: Month 6
Population: The PPS was defined as the subset of the FAS without any major protocol deviations. The FAS was defined as all participants randomized and who received an investigational product with at least one post-baseline effectiveness assessment (that is WSRS, blind evaluator's GAIS or participant's GAIS assessment).
Measure: Number; unit: Percentage of NLFs
Arm/Group | Radiesse | Restylane
Number analyzed (Participants) | 171 | 171
Percentage of NLFs | 78.4 | 83.3
Statistical Analysis 1: Comparison: Radiesse vs Restylane; Test type: Non-Inferiority — Non-inferiority margin, delta = 15%. The two-sided 95% CI for the differences between percentages was constructed using the Newcombe's recommended method; Difference in Percentage = -4.9, 95% CI 2-sided [-9.8 to -0.3]

ADVERSE EVENTS:
Time Frame: Baseline up to Month 12
Description: The investigator asked the participant for adverse events (AEs) systematically at each visit. The SES was used for AE assessment. The SES was defined as all participants who received an investigational product.
  As all participants received Radiesse in either of the two nasolabial folds and Restylane in the respective other, adverse events are reported in a combined group.
Arm/Group | Radiesse and Restylane
All-Cause Mortality (participants affected / at risk) | 0/176
Serious Adverse Events (participants affected / at risk) | 4/176
Other Adverse Events (participants affected / at risk) | 56/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiesse and Restylane (N=176)
Cervical dysplasia (Reproductive system and breast disorders) | 1
Endometrial thickening (Reproductive system and breast disorders) | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Radiesse and Restylane (N=176)
Urinary tract infection (Infections and infestations) | 16
Upper respiratory tract infection (Infections and infestations) | 11
Viral upper respiratory tract infection (Infections and infestations) | 10
Injection site nodule (General disorders) | 14 — 8 (4.5%) participants experienced this event at the Radiesse injection site, 9 (5.1%) at the Restylane injection site.
Hyperlipidaemia (Metabolism and nutrition disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the investigator will consider these doubts in the publication as long as the scientific neutrality is not affected.

DOCUMENTS (2):
  • Study Protocol (2018-07-27): https://cdn.clinicaltrials.gov/large-docs/57/NCT03282357/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT03282357/SAP_001.pdf